CLINICAL TRIAL: NCT03795441
Title: Open Label, Single Arm Phase 1 Study to Evaluate the Shedding, Biodistribution, Safety and Immunogenicity of Ad26.RSV.preF Vaccine in Adults
Brief Title: A Shedding Study of Adenovirus Serotype 26 Based Respiratory Syncytial Virus Pre-fusion F Protein (Ad26.RSV.preF) Vaccine in Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CR108554; 2018-003261-34 (EudraCT Number); VAC18193RSV1005 (Other: Janssen Vaccines & Prevention B.V.)
Record Dates: First submitted 2019-01-04; First posted 2019-01-07 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ad26.RSV.preF (Experimental): Participants will receive one intramuscular injection of an adenovirus serotype 26- based vaccine encoding for the respiratory syncytial virus pre-fusion F protein (Ad26.RSV.preF) on Day 1.
  Interventions: Biological: Ad26.RSV.preF

INTERVENTIONS:
Biological: Ad26.RSV.preF — Ad26.RSV.preF will be administered as intramuscular injection on Day 1.
  Other Names: JNJ-64400141

SUMMARY:
The purpose of this study is to assess the shedding and kinetics of the Adenovirus Serotype 26 Based Respiratory Syncytial Virus Pre-fusion F Protein (Ad26.RSV.preF) vaccine after one intramuscular injection of Ad26.RSV.preF in adults.

ELIGIBILITY:
Inclusion Criteria:

* In the investigator's clinical judgment, participant must be in good or stable health. Participants may have underlying illnesses such as hypertension, Type 2 diabetes mellitus, hyperlipoproteinemia, or hypothyroidism, as long as their symptoms and signs are medically controlled. If they are on medication for a condition, the medication dose must have been stable for at least 12 weeks preceding vaccination and expected to remain stable for the duration of the study. Participants will be included on the basis of physical examination, medical history, vital signs measurement and 12-lead electrocardiogram (ECG; for participants greater than [>] 65 years of age only) performed at screening
* Contraceptive use by women should be consistent with local regulations regarding the use of contraceptive methods for participants in clinical studies
* All women of childbearing potential must have a negative highly sensitive serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test at screening and a negative urine beta-hCG pregnancy test immediately prior to study vaccine administration
* From the time of vaccination through 3 months after vaccination, participant agrees not to donate blood
* Participant must be willing to provide verifiable identification, have means to be contacted and to contact the investigator during the study

Exclusion Criteria:

* Participant has a serious chronic disorder, including severe chronic obstructive pulmonary disease or clinically significant congestive heart failure, requirement for supplemental oxygen, end-stage renal disease with or without dialysis, clinically unstable cardiac disease, Alzheimer's disease, or has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (eg, compromise well-being) or that could prevent, limit, or confound the protocol-specified assessments
* Per medical history, participant has chronic active hepatitis B or hepatitis C infection
* Participant has received an investigational drug or used an invasive investigational medical device within 30 days or received an investigational vaccine within 6 months before the planned administration of study vaccine or is currently enrolled or plans to participate in another investigational study during the course of this study
* Participant has received treatment with immunoglobulin in the 2 months, or blood products in the 4 months before the planned administration of study vaccine or has any plans to receive such treatment during the study
* Participant has received any RSV vaccine in any previous RSV vaccine study at any time prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-07-28 (Actual); Study Completion 2019-07-28 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Presence of Ad26.RSV.preF (shedding) as Assessed by qPCR | Up to Day 183
  Percentage of Participants with presence of Ad26.RSV.preF in the adhesive bandage covering the injection site, the injection site area, nares (mid-turbinate), throat, rectum, urine, semen and blood, will be assessed by Quantitative Polymerase Chain Reaction (qPCR). Percentage of participants with presence of Ad26.RSV.preF (shedding) will be assessed.

SECONDARY OUTCOMES:
Number of Participants with Serious Adverse Events (SAEs) | First vaccination (Day 1) to the end of the study (Day 183)
  Number of participants with SAEs will be evaluated. An SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life threatening experience, is a congenital anomaly/birth defect, is suspected transmission of any infectious agent via a medicinal product, is medically important, and may jeopardize participant or may require medical or surgical intervention to prevent one of the outcomes listed above.
Number of Participants with Solicited Local and Systemic Adverse Events (AEs) After Vaccination | 7 days after vaccination (Day 1 up to Day 7)
  Number of participants with solicited local and systemic AEs will be evaluated. Solicited local AEs (erythema, swelling/induration, and pain/tenderness at the injection site) and solicited systemic AEs (fatigue, headache, myalgia, arthralgia, chills, nausea, and fever) will be noted in the participant diary through the 7 days post-vaccination. Local and systemic AEs will be graded according to severity as mild (Grade 1), moderate (Grade 2), severe (Grade 3) and potentially life threatening (Grade 4).
Number of Participants with Unsolicited AEs as a Measure of Safety | Day 1 Up to Day 28
  Number of participants with unsolicited AEs will be evaluated. An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non investigational) product, and it does not necessarily have a causal relationship with the intervention, therefore an AE can be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non investigational) product, whether or not related to that medicinal (investigational or non investigational) product. Unsolicited AEs will include all AEs for which the participant is specifically not questioned in the participant diary. Unsolicited AEs will be graded according to severity as mild (Grade 1), moderate (Grade 2), severe (Grade 3) and potentially life threatening (Grade 4).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency